CLINICAL TRIAL: NCT00088738
Title: Evaluation of Substance P Neurotransmission in Panic Disorder by PET Imaging of NK1 Receptors With [18F] SPA-RQ
Brief Title: Evaluation of Substance P Neurotransmission in Panic Disorder by PET Imaging of NK1 Receptors With [18F]SPA-RQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040189; 04-M-0189
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-09-10

CONDITIONS: Panic Disorder; Healthy
Keywords: Tachykinin; Anxiety; Neuroreceptor; Internalization; Carbon Dioxide; Healthy Volunteer; HV; Panic Disorder
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders | interventions — (2-fluoromethoxy-5-(5-trifluoromethyltetrazol-1-yl)benzyl)(2-phenylpiperidin-3-yl)amine

INTERVENTIONS:
Drug: [18F] SPA-RQ

SUMMARY:
This study is designed to observe the effects of a panic attack in patients with panic disorders and to demonstrate the involvement of Substance P in panic disorder, and thereby, further our understanding of its role in this illness. We will measure levels of Substance P in the brain by obtaining pictures of the brain using PET and MRI....

DETAILED DESCRIPTION:
The involvement of Substance P (SP) in depression and anxiety has been credibly demonstrated in a recent clinical trial. Although the precise physiological activation mechanism of the SP system is not yet known, the likelihood of exaggerated SP pathway activity in the pathogenesis of anxiety is supported in numerous animal studies that illustrate the anxiogenic, and anxiolytic effects of SP and SP antagonists (SPAs), respectively. Studies have further shown that SP release occurs in response to noxious, or aversive stimulation. SP stimulates NK1 receptors that then undergo endocytosis (i.e., internalization) resulting in a decrease in number of NK1 receptors on the cell surface. NK1 receptor quantification before, and after an aversive event, provides a dynamic measurement of SP neurotransmission.

In this protocol, we will use a new PET ligand that has demonstrated ability to serve as an NK1 receptor antagonist, [18F]SPA-RQ ( [18F]-labeled Substance P Antagonist Receptor Quantifier). Using this tracer, we will: 1.) quantify NK1 binding parameters and determine the reliability and reproducibility of these measures in 10 healthy controls, 2.) we will look for regional differences in NK1 receptor binding in 10 patients with panic disorder (PD) versus 10 normal controls, and 3.) We will perform a single-blind, placebo-controlled study to evaluate NK1 receptor binding in PD patients and controls following either saline or doxapram infusion, which is a respiratory stimulant, in 20 patients with panic disorder (PD) versus 20 normal controls. Doxapram acts on both peripheral and medullary chemoreceptors to increase the rate and depth of breathing. It appears to be a potent and specific panicogenic agent, triggering panic attacks. The majority of PD patients, but not controls, are expected to experience a panic attack (aversive event) following the doxapram infusion. Comparison of pre-panic and post-panic NK1 receptor binding in PD patients will provide an estimate of SP release. The goal of the present study is to demonstrate the involvement of SP in panic disorder, and thereby, further our understanding of its role in the psychopathology of this illness.

ELIGIBILITY:
* INCLUSION CRITERIA: (Phase 1) Whole Body Imaging
* Healthy Adults ages 18-50

EXCLUSION CRITERIA (Phase 1) Whole Body Imaging

* History of psychiatric disease, substance dependence or traumatic brain injury, severe systemic disease, poor vision or hearing
* History of substance abuse within 6 months
* Abnormal laboratory tests, including HIV test
* Any prior participation in other research protocols involving radiation exposure within the past year
* Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits. Limits: A total effective dose 2.5 rem in a year and 2.5 rad per year to the lens of the eyes, gonads and blood-forming organs; and 7.5 rad annually for all other organs.
* Pregnancy and Breast Feeding.
* Positive HIV test

INCLUSION CRITERIA: (Phase 2) Kinetic

* Ages 18-50
* Male or Female
* Informed consent given
* Subjects who regularly consume caffeinated beverages.

EXCLUSION CRITERIA: (Phase 2) Kinetic

* DSM-IV Axis I diagnostic criteria such as history of, or current Dx ADHD, mood/anxiety disorder, alcohol or psychoactive substance abuse/dependence
* Psychotropic medication or other drugs that may cross the blood brain barrier
* Traumatic brain injury, severe systemic disease
* Abnormal MRI other than minor atrophy
* Abnormal laboratory tests, including HIV test
* Claustrophobia
* Pregnancy or breast feeding
* Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits. Limits: A total effective dose or 5.0 rem in a year
* Any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.)
* Single radial and ulnar arterial circulation
* Individuals who recently donated blood
* Unable to lay on one's back for PET/MRI scans
* Novocaine allergy
* Positive HIV test

INCLUSION CRITERIA: (Phase 3A) Challenge

For Patients:

* Ages 18-65.
* DSM IV criteria for Panic Disorder
* Informed consent given.
* Subjects who regularly consume caffeinated beverages.

For Controls:

* Ages 18-65.
* Informed consent given.
* Subjects who regularly consume caffeinated beverages.

EXCLUSION CRITERIA: (Phase 3A) Challenge

For Patients and Controls:

* Current diagnosis of substance abuse or dependence
* History of substance dependence
* Psychotropic medication in last 3 weeks (8 weeks for fluoxetine/Prozac) except for benzodiazepene during PET or MRI scans
* Abnormal MRI other than minor atrophy
* Abnormal laboratory tests, including HIV test
* Pulmonary disease (e.g. COPD, asthma)
* Claustrophobia
* History of hypertension, coronary artery disease and subjects who are taking sympathomimetic medications
* Pregnancy or breastfeeding
* Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits. Limits: A total effective dose or 5.0 rem in a year
* Unable to lay on one's back for PET/MRI scans
* Any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.)

INCLUSION CRITERIA: (Phase 3B) Comparative

For Patients:

* Ages 18-65.
* DSM IV criteria for Panic Disorder
* Informed consent given.
* Subjects who regularly consume caffeinated beverages.

For Controls:

* Ages 18-65.
* Informed consent given.
* Subjects who regularly consume caffeinated beverages.

EXCLUSION CRITERIA: (Phase 3B) Comparative

For Patients and Controls:

* Current diagnosis of substance abuse or dependence
* History of substance dependence
* Psychotropic medication in last 3 weeks (8 weeks for fluoxetine/Prozac) except for benzodiazepene during PET or MRI scans
* Abnormal MRI other than minor atrophy
* Abnormal laboratory tests, including HIV test
* Pulmonary disease (e.g. COPD)
* Claustrophobia
* History of hypertension, coronary artery disease and subjects who are taking sympathomimetic medications
* Pregnancy or breastfeeding
* Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits. Limits: A total effective dose or 5.0 rem in a year
* Unable to lay on one's back for PET/MRI scans
* Any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2004-07-27; Study Completion 2008-09-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kramer MS, Cutler N, Feighner J, Shrivastava R, Carman J, Sramek JJ, Reines SA, Liu G, Snavely D, Wyatt-Knowles E, Hale JJ, Mills SG, MacCoss M, Swain CJ, Harrison T, Hill RG, Hefti F, Scolnick EM, Cascieri MA, Chicchi GG, Sadowski S, Williams AR, Hewson L, Smith D, Carlson EJ, Hargreaves RJ, Rupniak NM. Distinct mechanism for antidepressant activity by blockade of central substance P receptors. Science. 1998 Sep 11;281(5383):1640-5. doi: 10.1126/science.281.5383.1640. PMID 9733503
- [Background] Stockmeier CA, Shi X, Konick L, Overholser JC, Jurjus G, Meltzer HY, Friedman L, Blier P, Rajkowska G. Neurokinin-1 receptors are decreased in major depressive disorder. Neuroreport. 2002 Jul 2;13(9):1223-7. doi: 10.1097/00001756-200207020-00031. PMID 12151774
- [Background] Deguchi K, Antalffy BA, Twohill LJ, Chakraborty S, Glaze DG, Armstrong DD. Substance P immunoreactivity in Rett syndrome. Pediatr Neurol. 2000 Apr;22(4):259-66. doi: 10.1016/s0887-8994(00)00120-x. PMID 10788742